CLINICAL TRIAL: NCT06417814
Title: A Phase III, Open-label, Sponsor-blind, Randomized Study of Dato-DXd With or Without Osimertinib Versus Platinum-based Doublet Chemotherapy for Participants With EGFR-mutated Locally Advanced or Metastatic Non-small Cell Lung Cancer Whose Disease Has Progressed on Prior Osimertinib Treatment (TROPION-Lung15)
Brief Title: A Study to Investigate the Efficacy and Safety of Dato-DXd With or Without Osimertinib Compared With Platinum Based Doublet Chemotherapy in Participants With EGFR-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: TROPION-Lung15
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D516KC00001; 2024-511362-37-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: Epidermal growth factor receptor gene mutation; Standard of Care; Locally, advanced carcinoma; Metastatic carcinoma; Non-small cell lung cancer; Dato-dxd; Datopotamab deruxtecan; Osimertinib; Tagrisso; Pemetrexed; Carboplatin; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — osimertinib; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Dato-DXd + Osimertinib Combination Therapy (Experimental): Participants will receive Dato-DXd 6 milligrams per kilogram (mg/kg) as intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of every 21-day cycle, and osimertinib 80 milligrams (mg) once daily (QD) orally, until RECIST v1.1-defined radiological progression by investigator, unacceptable toxicity, or other discontinuation criterion is met.
  Interventions: Drug: Dato-DXd; Drug: Osimertinib
- Group 2: Dato-DXd Monotherapy (Experimental): Participants will receive Dato-DXd 6 mg/kg as IV infusion Q3W on Day 1 of every 21-day cycle, until RECIST v1.1-defined radiological progression by investigator, unacceptable toxicity, or other discontinuation criterion is met.
  Interventions: Drug: Dato-DXd
- Group 3: Platinum-based Doublet Chemotherapy (Experimental): Participants will receive pemetrexed 500 milligrams per meter square (mg/m2) in combination with carboplatin (AUC5) or cisplatin 75 mg/m2 as IV infusion Q3W for 4 cycles followed by pemetrexed maintenance 500 mg/m2 as IV infusion Q3W, until RECIST v1.1-defined radiological progression by investigator, unacceptable toxicity, or another discontinuation criterion is met.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Dato-DXd — Dato-DXd will be administered as IV infusion.
  Other Names: DS-1062a
  Arms: Group 1: Dato-DXd + Osimertinib Combination Therapy; Group 2: Dato-DXd Monotherapy
Drug: Osimertinib — Osimertinib will be administered orally.
  Other Names: Tagrisso; AZD9291
  Arms: Group 1: Dato-DXd + Osimertinib Combination Therapy
Drug: Pemetrexed — Pemetrexed will be administered as IV infusion.
  Arms: Group 3: Platinum-based Doublet Chemotherapy
Drug: Carboplatin — Carboplatin will be administered as IV infusion.
  Arms: Group 3: Platinum-based Doublet Chemotherapy
Drug: Cisplatin — Cisplatin will be administered as IV infusion.
  Arms: Group 3: Platinum-based Doublet Chemotherapy

SUMMARY:
This study will assess the effect of Dato-DXd in combination with osimertinib or Dato-DXd monotherapy versus platinum-based doublet chemotherapy in terms of progression-free survival (PFS).

DETAILED DESCRIPTION:
This is a Phase III, open-label, 3-arm, multicenter study assessing the effects of Dato-DXd in combination with osimertinib or Dato-DXd monotherapy versus platinum-based doublet chemotherapy in participants with epidermal growth factor receptor gene mutation (EGFRm) locally advanced or metastatic non-small cell lung cancer (NSCLC) whose disease has progressed on prior osimertinib treatment.

Participants will be randomized in a 1:1:1 ratio to one of the following intervention groups:

1. Dato-DXd + osimertinib combination therapy
2. Dato-DXd monotherapy
3. Platinum-based doublet chemotherapy

Participants will receive study intervention until Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) -defined radiological progression by the investigator, unacceptable toxicity, or other discontinuation criterion is met.

After study intervention discontinuation, all participants will undergo an end of treatment (EoT) visit within 35 days of discontinuation and will be followed up for safety assessments 28 (+ 7) days after their last dose of study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-squamous NSCLC.
* Must have evidence of documented pre-existing EGFRm information (EGFRm known to be associated with (epidermal growth factor receptor [EGFR] tyrosine kinase inhibitor [TKis] sensitivity [Ex19del, L858R, G719X, S768I, or L861Q], either alone or in combination with other EGFR mutations, which may include T790M).
* Documented extra-cranial radiologic progression on prior osimertinib monotherapy (as most recent line of treatment) in the adjuvant, locally advanced, or metastatic setting.
* Less than or equal to (<=2) prior lines of EGFR TKIs (osimertinib is the only permitted prior third generation EGFR TKI).
* At least one lesion, not previously irradiated, that qualifies as a RECIST v1.1 TL at baseline and can be accurately measured at baseline.
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow reserve and organ function within 7 days before randomization.

Exclusion Criteria:

* Use of chemotherapy, vascular endothelial growth factor inhibitor, immunotherapy or any anti-cancer therapy in the metastatic setting. Platinum-based chemotherapy in non-metastatic setting within 12 months prior to randomization.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 2 years before the first dose of study intervention.
* Any evidence of severe or uncontrolled systemic diseases, including, but not limited to active bleeding diseases, active infection, active ILD/pneumonitis, cardiac disease.
* Has significant third-space fluid retention (example [eg.], ascites or pleural effusion) as judged by the investigator and is not amenable for required repeated drainage.
* History of non-infectious ILD/pneumonitis including radiation pneumonitis that required steroids or drug-induced ILD, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
* Has severe pulmonary function compromise resulting from intercurrent pulmonary illnesses.
* Unstable spinal cord compression and/or unstable brain metastases.
* Participants with symptomatic brain metastases (including leptomeningeal involvement).
* Clinically significant corneal disease.
* Uncontrolled infection requiring systemic antibiotics, antivirals, or antifungals, suspected infections or inability to rule out infections. Use of systemic antibiotics within 14 days of randomization.
* Has known human immunodeficiency virus (HIV) infection that is not well controlled.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-27 (Estimated)

PRIMARY OUTCOMES:
Progression free Survival (PFS) | Up to 2.5 years
  PFS is defined as the time from randomization to Blinded Independent Central Review (BICR)-assessed progression using RECIST v1.1 or death due to any cause, regardless of whether the participant withdraws from study therapy, receives other anti-cancer therapy, or clinical progression.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3.5 years
  OS is defined as time from randomization until the date of death due to any cause.
Central Nervous System Progression-free Survival (CNS PFS) | Up to 2.5 years
  CNS PFS is defined as the time from randomization to BICR confirmed progression in the CNS or death due to any cause, regardless of whether the participant withdraws from study therapy, receives other anti-cancer therapy, or clinically progresses prior to BICR confirmed CNS modified RECIST v1.1 progression.
Objective Response Rate (ORR) | Up to 2.5 years
  ORR is defined as the percentage of participants who have a confirmed complete response (CR) or confirmed partial response (PR), as determined by BICR per RECIST v1.1.
Duration of Response (DoR) | Up to 2.5 years
  DoR is defined as the time from the date of first documented response until date of documented progression per RECIST v1.1, as assessed by BICR or death due to any cause.
Progression-free Survival-2 (PFS-2) | Up to 3.5 years
  PFS2 is defined as the time from randomization to the earliest of the progression event (following the initial investigator assessed progression), after first subsequent therapy, or death.
Objective Response Rate (ORR) Using CNS Modified RECIST v1.1 | Up to 2.5 years
  ORR is defined as the percentage of participants who have a confirmed CR or confirmed PR, using CNS modified RECIST v1.1.
Duration of Response (DoR) Using CNS Modified RECIST v1.1 | Up to 2.5 years
  DoR is defined as the time from the date of first documented response until date of documented progression or death due to any cause using CNS modified RECIST v1.1.
Time to Deterioration in Pulmonary Symptoms | Up to 3.5 years
  Time to deterioration (in pulmonary symptoms [dyspnea, cough, and chest pain]) is defined as the time from randomization until the date of deterioration. Deterioration is defined as change from baseline that reaches a meaningful change threshold.
Time to Deterioration in Physical Functioning | Up to 3.5 years
  Time to deterioration in physical functioning as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function short form 8c will be evaluated. Time to deterioration (in physical functionating) is defined as the time from randomization until the date of deterioration. Deterioration is defined as change from baseline that reaches a meaningful change threshold.
Time to Deterioration in Global Health Status (GHS)/Quality of Life (QoL) | Up to 3.5 years
  Time to deterioration in GHS/QoL as measured by the GHS/QoL scale from EORTC IL172 will be reported. Time to deterioration (in GHS/QoL) is defined as the time from randomization until the date of deterioration. Deterioration is defined as change from baseline that reaches a meaningful change threshold.
Pharmacokinetics (PK) of Dato-DXd | Up to 3.5 years
  Concentration of Dato-DXd, total anti-TROP2 antibody and DXd in plasma.
Immunogenicity of Dato-DXd | Up to 3.5 years
  Presence of antidrug antibody (ADAs) for Dato-DXd (confirmatory results: positive or negative, titers).

CONTACTS AND LOCATIONS:
Locations (246):
- United States (31):
  - Research Site, Fayetteville, Arkansas
  - Research Site, Duarte, California
  - Research Site, Fountain Valley, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Athens, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Morristown, New Jersey
  - Research Site, Northfield, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Maumee, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
- Australia (10):
  - Research Site, Fitzroy
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Liverpool
  - Research Site, Nedlands
  - Research Site, Port Macquarie
  - Research Site, St Leonards
  - Research Site, Westmead
  - Research Site, Woodville
  - Research Site, Woolloongabba
- Belgium (9):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Jette
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Roeselare
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Betim
  - Research Site, Blumenau
  - Research Site, Florianópolis
  - Research Site, Itajaí
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Brampton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (26):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Deyang
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Huaian
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Luoyang
  - Research Site, Luzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- France (14):
  - Research Site, Angers
  - Research Site, Avignon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Quimper
  - Research Site, Toulon Armees
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Berlin
  - Research Site, Berlin-Zehlendorf
  - Research Site, Bonn
  - Research Site, Essen
  - Research Site, Georgsmarienhütte
  - Research Site, Giessen
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kempten
  - Research Site, Löwenstein
  - Research Site, Nuremberg
  - Research Site, Oldenburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (14):
  - Research Site, Amravati
  - Research Site, Bhubaneswar
  - Research Site, Hyderabad
  - Research Site, Kolhāpur
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, Namakkal
  - Research Site, Pune
  - Research Site, Raipur
  - Research Site, Rajasthan
  - Research Site, Ranchi
  - Research Site, Thane
  - Research Site, Trivandrum
  - Research Site, Varanasi
- Israel (7):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (12):
  - Research Site, Bari
  - Research Site, Milan
  - Research Site, Misterbianco
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Verona
- Japan (20):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Iruma-Gun
  - Research Site, Iwakuni-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ōsaka-sayama
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
  - Research Site, Utsunomiya
  - Research Site, Wakayama
  - Research Site, Yokohama
- Malaysia (8):
  - Research Site, Alor Star
  - Research Site, Cheras
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
  - Research Site, Perai
  - Research Site, Petaling Jaya
- Netherlands (4):
  - Research Site, Amersfoort
  - Research Site, Harderwijk
  - Research Site, Rotterdam
  - Research Site, Zutphen
- Philippines (6):
  - Research Site, Bacolod
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Manila
  - Research Site, Quezon
  - Research Site, San Juan City
- Poland (5):
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
- Portugal (4):
  - Research Site, Braga
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
- Research Site, Craiova, Romania
- Research Site, Singapore, Singapore
- South Korea (7):
  - Research Site, Busan
  - Research Site, Chungcheongbuk-do
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (16):
  - Research Site, A Coruña
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Santiago de Compostela-Coruña
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Pathum Thani
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Middlesbrough
- Research Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
  For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tan DS, Nadal E, Cheema P, Wu YL, Ahn MJ, Tanizaki J, Grainger E, Nizialek E, Forcina A, van der Gronde T, Yu HA. TROPION-Lung15: a randomized phase III study of osimertinib combined with datopotamab deruxtecan (Dato-DXd) or Dato-DXd alone versus platinum-doublet chemotherapy in patients with EGFR-mutated advanced non-small cell lung cancer and whose disease has progressed on prior osimertinib. Ther Adv Med Oncol. 2025 Dec 23;17:17588359251385410. doi: 10.1177/17588359251385410. eCollection 2025. PMID 41466843